CLINICAL TRIAL: NCT06914063
Title: Assessing Patient Comfort, Anxiety, and Satisfaction During Cycloplegic Refraction: Comparing Conventional Drops With Rapid-Onset Cycloplegics
Brief Title: Assessing Patient Comfort, Anxiety, and Satisfaction During CR Comparing Conventional Drops With ROC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/813
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cycloplegic Paralysis of Accommodation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid-Onset Cycloplegic Drops (Experimental)
  Interventions: Combination Product: Rapid-Onset Cycloplegic Drops
- Conventional Cycloplegic Drops (Active Comparator)
  Interventions: Diagnostic Test: Conventional Cycloplegic Drops

INTERVENTIONS:
Combination Product: Rapid-Onset Cycloplegic Drops — Rapid-Onset Cycloplegic Drops (e.g., tropicamide with phenylephrine) to assess patient comfort, anxiety, and satisfaction with quicker onset and shorter duration.
  Arms: Rapid-Onset Cycloplegic Drops
Diagnostic Test: Conventional Cycloplegic Drops — Conventional Cycloplegic Drops (e.g., cyclopentolate) to provide a baseline for comparison with the rapid-onset treatment.
  Arms: Conventional Cycloplegic Drops

SUMMARY:
This study aims to compare the efficacy of conventional cycloplegic agents, such as cyclopentolate, with rapid-onset cycloplegics, like a combination of tropicamide and phenylephrine, in reducing patient anxiety and discomfort during cycloplegic refraction. Cycloplegic refraction is an essential procedure for diagnosing refractive errors, particularly in children, by temporarily paralyzing the ciliary muscle to inhibit accommodation. While cyclopentolate has a relatively quick onset, tropicamide is preferred due to its faster onset and shorter duration. Despite its advantages, concerns about patient discomfort and anxiety during the procedure remain, especially in pediatric populations.

DETAILED DESCRIPTION:
The study will involve participants aged 3-16 years, with no significant refractive error or ocular pathologies. Patients will be randomly assigned to receive either cyclopentolate or tropicamide with phenylephrine. The primary outcomes include patient comfort, anxiety levels, satisfaction, and procedure time. Discomfort and anxiety will be measured using questionnaires such as the Visual Analog Scale for Comfort and the State-Trait Anxiety Inventory. The study will help determine if rapid-onset cycloplegic provide a better patient experience by reducing discomfort and anxiety. By evaluating these factors, the research seeks to improve clinical practices in optometry and ophthalmology, particularly in pediatric eye examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10-20years.
* Both Male and Female
* Healthy participants with no abnormalities detected in anterior segment structures or fundus examination using slit-lamp biomicroscopy and a 90-diopter lens.
* No significant refractive error (within the range of ±1 diopter in spherical equivalent).

Exclusion Criteria:

* History of severe allergic reactions or adverse effects to cycloplegic agents
* Severe anxiety, panic disorders, or other psychological conditions that may interfere with reporting the experience accurately.
* Uncontrolled systemic diseases (e.g., uncontrolled diabetes or cardiovascular conditions) that may impact the response to cycloplegic agents.
* Recent ocular surgery (e.g., LASIK, cataract surgery) or eye trauma affecting refraction accuracy or comfort.
* Presence or history of any intraocular diseases, including glaucoma, uveitis, and retinal disorders.
* Systemic disorders such as hypertension, cardiovascular disease, or respiratory disease.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  The Visual Analogue Scale (VAS) score is a pain measurement tool where patients mark a point on a 10 cm line representing their pain intensity, with the distance from "no pain" measured in millimeters (0-100), indicating pain intensity
State-Trait Anxiety Inventory (STAI) | 12 Months
  The State-Trait Anxiety Inventory (STAI) is a 40-item self-report questionnaire measuring anxiety, divided into 20 items for state anxiety (how one feels now) and 20 for trait anxiety (how one generally feels). Each item is scored on a 4-point Likert scale, with higher scores indicating greater anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shifa trust eye Hospital, Sukkur, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No